CLINICAL TRIAL: NCT02827981
Title: Retrospective Study on the Evaluation of Intra-disc Infiltration in the Active Disc Disease
Acronym: MODIC
Status: Withdrawn | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: MODIC
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2016-06

CONDITIONS: Disc Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Active discopathies or MODIC 1, are a diagnostic entity discovery with the contribution of MRI in which the first cases were described by Dr. Michael MODIC in 1988. It is characterized by a vertebral bone edema secondary to active discarthrose. Its prevalence is estimated at 6% of the general population and up to 40% of the CLBP according to studies. Following the discovery of this recent diagnostic entity, responsible for low back pain, the question of its management is debate in the medical community. Early studies demonstrate the effectiveness of corticosteroid injections in intra-disc. Other works, most recent, suggest the contrary, infectious, incriminating a pathogenic role of certain bacteria such as Propionibacterium acness or Corynebacterium propinquum recommending, in contrast, treatment with prolonged antibiotic therapy. This study will aim to assess the effectiveness of intra-disc infiltration GHPSJ carried out between 2007 and 2014. The innovation of our work will be to assess these infiltrations in various subgroups such as patients with a previous surgery of the spine or a history of scoliosis or spondylolisthesis.

DETAILED DESCRIPTION:
1. Primary objective:

   Evaluate the effectiveness of intra-disc infiltrations conducted in the rheumatology department of pain in the active disc disease.
2. Secondary objectives:

   * Evaluate the duration of the benefit on pain caused by gesture
   * Assess the impact of the gesture on NSAIDs and / or analgesics
   * Analysis of different subgroups (antecedent of surgery, spondylolisthesis, scoliosis) Inclusion / non-inclusion: Patients older than 18 who were hospitalized between 2007 and 2014 in the Rheumatology Department for intradiscal infiltration.

Methodology: A retrospective, single-center, non-interventional Study duration: 6 months Acquisition of data: demographic data, data on the disc disease, data on the assessment of pain, the effectiveness of infiltration of analgesics and / or NSAIDs, or need infiltration surgery for the gesture.

Supports: patient questionnaire report hospital, medical, Excel grid of data collection), analysis (statistic: local management) Anonymised data in the Excel spreadsheet Development of the study: Data collection, statistical analysis, literature review Retrospective study based on recovering data regarding efficacy of infiltrative gesture that some patient was performed in 2007, with possibility of bias on the recovery of data in view of the age of the gesture for some patients.

An analysis of each folder from the hospital report will be carried out in parallel in order to compare the data collected by the questionnaire with the reporting. The sending of questionnaires and letters will be performed by the service attaches where a pre-stamped letter. The address of the patients will be that recorded in the base DxCare.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged > 18yo
* Hospitalization between 2007 and 2014 in the Rheumatology Department for intradiscal infiltration

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized between 2007 and 2014 in the Rheumatology Department for intradiscal infiltration.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pain Scores on visual Analogue Scale | Day1, Before and after Intra-disc Infiltration
  Change From Baseline in Pain Scores on the Visual Analog Scale at 6 Weeks

SECONDARY OUTCOMES:
Amount of analgesic taken | Day1

CONTACTS AND LOCATIONS:
Overall Officials: ISRAEL Jonathan, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe hospitalier Paris Saint-Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided